CLINICAL TRIAL: NCT04228081
Title: The Development of a Rapid and Accurate Method for Detecting and Susceptibility Testing of Bacteria Causing Urinary Tract Infection Using a Metabolomic Platform
Brief Title: MicroUDxTM: a Rapid Diagnostic Tool That Will Prevent Death and Disability From Common Infections
Acronym: MicroUDxTM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Ian Lewis, Assistant Professor, University of Calgary
Other Study IDs: REB19-00442
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Bacterial Urinary Tract Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — research samples will be stored in a equal volume of 100% methanol in a -80 freezer at the Diagnostic and Scientific Centre or at the Lewis Lab in Biological Sciences U of C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UTI Positive: In phase I of the study testing residual urine samples the aim is to include at least 50 positive samples from each bacterial species known to be commonly associated with urinary tract infections. We selected 2000 positive urines to enable capturing enough of these organisms in the development process.
  For phase II of the study, the same number of positive samples in order to include all common species causing urinary tract infection. The number of negative samples included is reduced to 1000.
  Phase 3 - approximately one third of all urine sample submitted will be positive for a uropathogen. Sample size of 3000 we expect 1000 these to be culture positive. We expect most uropathogens occurring at a frequency of 5% or more will be included with sufficient numbers in the validation process.
- UTI Negative Control: 2000 negative urine samples are being run as controlled to ensure the false positivity rate is low.

SUMMARY:
Background & Rational:

Antibiotics are a major underpinning of modern medicine. The global rise of antimicrobial resistant (AMR) organisms is a serious world health problem. With few new antimicrobial drugs on the horizon, it is imperative that we develop novel approaches to extend the service life of our existing drugs. AMR is a complex problem that is being driven by a wide range of factors. More than half of the antibiotics prescribed have no medical benefit, and outpatient visits for uncomplicated urinary tract infections (UTIs) are a major contributor to this problem. Recent studies have shown that nearly half of people treated for UTIs receive the wrong frontline drug and in 75% of patients, the duration of therapy is inappropriate. Limitations in the current diagnostic technology make it impossible to identify UTI pathogens and measure their antibiotic sensitivities during the short out-patient clinical visits that are typical for most UTI patients. These circumstances result in the inappropriate use of stronger than necessary or inappropriate antimicrobials. The aim of this study is to develop and evaluate a system that can detect bacteria in urine and find the best antibiotic in under 4 hours, thus enabling a rapid diagnosis and use of the most appropriate and cost-effective antimicrobial agent for the agent detected.

DETAILED DESCRIPTION:
Testing done in this study will be performed either on bacterial isolates stored in the microbiology laboratory at the Diagnostic and Scientific Center in Calgary, or on up to one milliliter of residual urine sample submitted to the diagnostic laboratory with a request for urine culture and sensitivity. All urine cultures will be performed and reported in accordance with standards laboratory protocols. Research testing will only be done on residual sample once patient samples are processed or reported on for clinical purposes.

During the first phase of the study, metabolic biomarkers for uropathogens will be identified using mass spectrometry on sub-cultures of frozen isolates from the diagnostic microbiology laboratory. This will include at least 50 isolates each of uropathogens consisting of but not limited to Escherichia coli, Klebsiella oxytoca, Klebsiella pneumoniae, Enterobacter species, Proteus mirabilis, Citrobacter species, Staphylococcus aureus, Staphylococcus saprophyticus, Pseudomonas aeruginosa, Enterococcus species, and Candida species. Biomarkers that are present in greater than 95% of the isolates will subsequently be using the analysis of 2000 negative, and 2000 positive urine cultures. Compounds that are subsequently identified as high yield will be selected for carbon 13 labeling to service standards.

In phase II of the study, following the development of a biomarker enrichment device at the CMRF, a performance urinalysis of the device will be conducted using residual urine sample from 1000 negative and 2000 positive urine specimens as outlined above. The performance of the new device will be evaluated relative to standard cultures and urine liquid chromatography-mass spectrometry.

Following the creation of a sensitive and specific assay, a prospective study will be carried out at the diagnostic microbiology laboratory. 3000 sample submitted for urine culture will be process in parallel with the new device and standard microbiology procedures. Sensitivity, specificity and predictive value for each analyte compared to standard culture will be determined in this portion of the study. Cost calculations and performance characteristics including turnaround time of the new assay will be compared to that in the standard laboratory procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have not submitted urine samples will not be included as the samples are required for both standard testing and research. This would include patients who are being treated empirically by physicians.

Exclusion Criteria:

* Patient's who have not submitted urine samples for culture will not be included in study.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The majority of urine samples collected in Calgary coming from young healthy females with symptoms of cystitis or pyelonephritis. However, residual sample from any patient where a urine culture has been ordered could be included in the study if it falls within the time during which residual samples are being processed.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Assay ID Validation | 2 years
  In the validation phase of the study sensitivity, specificity and positive and negative predictive values for detecting significant bacteriuria using culture as the gold standard, These values will be calculated for the whole cohort as per standard definitions using statistical software (Analyse-it for Excel).

SECONDARY OUTCOMES:
Susceptibility - anti-microbial susceptibility of new assay versus standard laboratory methods | 2 years
  A secondary outcome variable will be the detection of antimicrobial susceptibility using the new assay will be the calculation of essential and categorical agreement, major, very major and minor errors between the new assay and standard laboratory methods as per standard laboratory definitions.
Turn-around-time to bacterial detection and susceptibility | 2 years
  Another secondary outcome will be the turn-around- time (TAT) to bacterial detection and availability of susceptibility results.

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Lewis, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No data will be made available to other researchers